CLINICAL TRIAL: NCT06252805
Title: Severe Prospective Observational Study of COPD in Catalonia
Brief Title: Severe Prospective Observational COPD Catalonia
Acronym: SPOCCAT
Status: Not yet recruiting | Type: Observational
Sponsor: Ferran Morell (Other)
Responsible Party: Sponsor-Investigator, Ferran Morell, president, Fundacio Catalana de Pneumologia
Organization: Fundacio Catalana de Pneumologia (Other)
Other Study IDs: FUC-SPOCCAT-2023-10
Record Dates: First submitted 2023-10-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Severe Chronic Obstructive Pulmonary Disease
Keywords: Severe COPD; Cohort; Catalonia; Prospective; Multicenter; 5 year follow-up; characterisation; COPD comorbidities; COPD phenotypes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPOCCAT: Severe Chronic Obstructive Pulmonary Disease patients in Catalonia

SUMMARY:
Multicenter observational study to characterize and follow-up a cohort of patients with severe chronic obstructive pulmonary disease (COPD) in Catalonia

DETAILED DESCRIPTION:
Creation of the first multicenter observational study in Catalonia to characterize and follow-up of patients with severe chronic obstructive pulmonary disease. The follow-up will be up to 5 years, with a first initial visit and control visits every year. All patients will be recruited from respiratory departments from major hospitals from Catalonia, a region with approximately 8 million inhabitants and a wide web of public hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: a signed and dated written informed consent prior to study participation
* Age: Subjects 35 years of age or order at visit 1.
* Severe COPD diagnosis: an established severe COPD defined by spirometry values:

  * A post-albuterol/salbutamol FEV1/FVC ratio of <0.70 at visit 1. FEV1: forced expiratory volume at one second FVC: forced vital capacity.
  * A post-bronchodilator FEV1 < 50% predicted normal
* Smoking history: ≥ 10 pack-years at visit 1
* Stable phase of the disease (not less than 4 weeks of stability prior visit 1)

Exclusion Criteria:

* Subjects not giving written informed consent.
* Subjects at risk of non-compliance, or unable to comply with the scheduled visits.
* Subjects affected mainly by another severe chronic respiratory disease that justifies the ventilatory alteration, for example pulmonary fibrosis or severe bronchiectasis
* Subjects with carcinoma that has not been in complete remission for at least 5 years.
* Subjects with α1-antitrypsin deficiency as the underlying cause of COPD

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD subjects from respiratory departments in Hospitals from Catalonia
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Cohort creation in Catalonia | Up to 5 years
  Creation of a long follow-up (5 years) cohort of severe COPD patients in Catalonia
Describe the demographic and clinical characteristics of patients with severe COPD in Catalonia. | Up to 5 years
  Identify the distribution of sex, age, severity of lung function impairment, treatment administered and comorbidities of severe COPD patients
Assess the natural history and prognosis of severe COPD | Up to 5 years
  Assess the decline in lung function, frequency and severity of exacerbations and survival over a period of 5 years

SECONDARY OUTCOMES:
Assess effect of the different treatments, both inhaled and non-inhaled, on the disease progression and according to the patient's phenotype. | Up to 5 years
  Compare the evolution in terms of decline in lung function, exacerbations and survival in patients treated with inhaled corticosteroids versus patients treated without inhaled corticosteroids
Impact of exacerbations and chronic bronchial infection on the evolution of COPD | Up to 5 years
  Compare the evolution in terms of decline in lung function, frequency and severity of exacerbations and survival according to the presence and severity of exacerbations and the presence of chronic bronchial infection during follow-up
Importance of comorbidities in the evolution of COPD | Up to 5 years
  Compare the evolution in terms of decline in lung function, frequency and severity of exacerbations and survival according to the presence and severity of different comorbidities and according to the scores on the Chrlson comorbidity index

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Almagro P, Soriano JB, Cabrera FJ, Boixeda R, Alonso-Ortiz MB, Barreiro B, Diez-Manglano J, Murio C, Heredia JL; Working Group on COPD, SpanishSociety of Internal Medicine*. Short- and medium-term prognosis in patients hospitalized for COPD exacerbation: the CODEX index. Chest. 2014 May;145(5):972-980. doi: 10.1378/chest.13-1328. PMID 24077342
- [Background] Fletcher C, Peto R. The natural history of chronic airflow obstruction. Br Med J. 1977 Jun 25;1(6077):1645-8. doi: 10.1136/bmj.1.6077.1645. PMID 871704
- [Background] Lokke A, Lange P, Scharling H, Fabricius P, Vestbo J. Developing COPD: a 25 year follow up study of the general population. Thorax. 2006 Nov;61(11):935-9. doi: 10.1136/thx.2006.062802. PMID 17071833
- [Background] Kohansal R, Martinez-Camblor P, Agusti A, Buist AS, Mannino DM, Soriano JB. The natural history of chronic airflow obstruction revisited: an analysis of the Framingham offspring cohort. Am J Respir Crit Care Med. 2009 Jul 1;180(1):3-10. doi: 10.1164/rccm.200901-0047OC. Epub 2009 Apr 2. PMID 19342411
- [Background] Vestbo J, Anderson W, Coxson HO, Crim C, Dawber F, Edwards L, Hagan G, Knobil K, Lomas DA, MacNee W, Silverman EK, Tal-Singer R; ECLIPSE investigators. Evaluation of COPD Longitudinally to Identify Predictive Surrogate End-points (ECLIPSE). Eur Respir J. 2008 Apr;31(4):869-73. doi: 10.1183/09031936.00111707. Epub 2008 Jan 23. PMID 18216052
- [Background] Garcia-Aymerich J, Gomez FP, Anto JM; en nombre del Grupo Investigador del Estudio PAC-COPD. [Phenotypic characterization and course of chronic obstructive pulmonary disease in the PAC-COPD Study: design and methods]. Arch Bronconeumol. 2009 Jan;45(1):4-11. doi: 10.1016/j.arbres.2008.03.001. Epub 2009 Jan 3. Spanish. PMID 19186292
- [Background] Regan EA, Hokanson JE, Murphy JR, Make B, Lynch DA, Beaty TH, Curran-Everett D, Silverman EK, Crapo JD. Genetic epidemiology of COPD (COPDGene) study design. COPD. 2010 Feb;7(1):32-43. doi: 10.3109/15412550903499522. PMID 20214461
- [Background] Makita H, Nasuhara Y, Nagai K, Ito Y, Hasegawa M, Betsuyaku T, Onodera Y, Hizawa N, Nishimura M; Hokkaido COPD Cohort Study Group. Characterisation of phenotypes based on severity of emphysema in chronic obstructive pulmonary disease. Thorax. 2007 Nov;62(11):932-7. doi: 10.1136/thx.2006.072777. Epub 2007 Jun 15. PMID 17573447
- [Background] Kunzli N, Ackermann-Liebrich U, Keller R, Perruchoud AP, Schindler C. Variability of FVC and FEV1 due to technician, team, device and subject in an eight centre study: three quality control studies in SAPALDIA. Swiss Study on Air Pollution and Lung Disease in Adults. Eur Respir J. 1995 Mar;8(3):371-6. doi: 10.1183/09031936.95.08030371. PMID 7789479
- [Background] Downs SH, Brandli O, Zellweger JP, Schindler C, Kunzli N, Gerbase MW, Burdet L, Bettschart R, Zemp E, Frey M, Keller R, Tschopp JM, Leuenberger P, Ackermann-Liebrich U; SAPALDIA team. Accelerated decline in lung function in smoking women with airway obstruction: SAPALDIA 2 cohort study. Respir Res. 2005 May 26;6(1):45. doi: 10.1186/1465-9921-6-45. PMID 15918902
- [Background] Lopez-Campos JL, Peces-Barba G, Soler-Cataluna JJ, Soriano JB, de Lucas Ramos P, de-Torres JP, Marin JM, Casanova C; en nombre del grupo de estudio CHAIN. Chronic obstructive pulmonary disease history assessment in Spain: a multidimensional chronic obstructive pulmonary disease evaluation. Study methods and organization. Arch Bronconeumol. 2012 Dec;48(12):453-9. doi: 10.1016/j.arbres.2012.05.006. Epub 2012 Jul 4. English, Spanish. PMID 22766419
- [Background] Calle Rubio M, Rodriguez Hermosa JL, de Torres JP, Marin JM, Martinez-Gonzalez C, Fuster A, Cosio BG, Peces-Barba G, Solanes I, Feu-Collado N, Lopez-Campos JL, Casanova C; CHAIN Study Investigators. COPD Clinical Control: predictors and long-term follow-up of the CHAIN cohort. Respir Res. 2021 Feb 4;22(1):36. doi: 10.1186/s12931-021-01633-y. PMID 33541356
- [Background] Chen CZ, Shih CY, Hsiue TR, Tsai SH, Liao XM, Yu CH, Yang SC, Wang JD. Life expectancy (LE) and loss-of-LE for patients with chronic obstructive pulmonary disease. Respir Med. 2020 Oct;172:106132. doi: 10.1016/j.rmed.2020.106132. Epub 2020 Aug 29. PMID 32905891
- [Result] Soriano JB, Alfageme I, Miravitlles M, de Lucas P, Soler-Cataluna JJ, Garcia-Rio F, Casanova C, Rodriguez Gonzalez-Moro JM, Cosio BG, Sanchez G, Ancochea J. Prevalence and Determinants of COPD in Spain: EPISCAN II. Arch Bronconeumol (Engl Ed). 2021 Jan;57(1):61-69. doi: 10.1016/j.arbres.2020.07.024. Epub 2020 Sep 17. English, Spanish. PMID 32950310
- See also: GOLD COPD 2023 report (GOLD: Global Initiative for Chronical Obstructive Lung Disease) — https://goldcopd.org/2023-gold-report-2
- See also: WHO (World Health Organization). The Top 10 causes ofr death — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death